CLINICAL TRIAL: NCT03688542
Title: Opportunities and Limits to Deprescribing in Nursing Homes:Quality Circle Deprescribing Module
Acronym: OLD-NH-QC-DeMo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anne Niquille (Other)
Responsible Party: Sponsor-Investigator, Anne Niquille, Dr, University of Geneva, Switzerland
Organization: University of Geneva, Switzerland (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: OLD-NH-QC-DeMo-2017
Record Dates: First submitted 2018-09-26; First posted 2018-09-28 (Actual); Results first posted 2021-04-21 (Actual); Last update posted 2021-04-21 (Actual); Status verified 2021-03

CONDITIONS: Polypharmacy; Inappropriate Prescribing
Keywords: Deprescribing; Inappropriate Medication; Nursing Homes

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Nursing Homes allocated to the Intervention arm will enact the Quality Circle Deprescribing Module and create a local deprescribing consensus and implementation strategy.
  Interventions: Other: Quality Circle Deprescribing Module
- Control (No Intervention): Nursing Homes allocated to the Control arm will not enact the intervention.

INTERVENTIONS:
Other: Quality Circle Deprescribing Module — The Quality Circle Deprescribing Module consist of a discussion bringing together nurses, physicians and responsible pharmacist to create a local deprescribing consensus for frequently used drug classes, as well as implementation strategies for the consensus..
  Arms: Intervention

SUMMARY:
Older people residing in nursing homes (NH) are frequently polymedicated and often prescribed potentially inappropriate medications. Deprescribing has been proposed as a way to reduce the number of drugs they receive and their exposure to harmful treatments.

The objectives of this study are 1) To evaluate the effect of a deprescribing-specific interdisciplinary quality circle module on the use of potentially inappropriate medication in nursing-home residents. 2) To determine the effective strategies to reach and implement deprescribing consensus resulting of said quality circle module.

ELIGIBILITY:
Inclusion Criteria:

Nursing homes taking part in the study must have

* a geriatric of psycho-geriatric mission;
* been part of their cantonal pharmaceutical assistance program for at least a year.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2017-09-25 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Bugnon, Prof, Study Director — University of Geneva
Locations (1):
- Centre de Pharamacie Communautaire, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mena S, Moullin JC, Schneider M, Niquille A. Implementation of interprofessional quality circles on deprescribing in Swiss nursing homes: an observational study. BMC Geriatr. 2023 Oct 3;23(1):620. doi: 10.1186/s12877-023-04335-w. PMID 37789286
- [Derived] Cateau D, Ballabeni P, Niquille A. Effects of an interprofessional deprescribing intervention in Swiss nursing homes: the Individual Deprescribing Intervention (IDeI) randomised controlled trial. BMC Geriatr. 2021 Nov 19;21(1):655. doi: 10.1186/s12877-021-02465-7. PMID 34798826
- [Derived] Cateau D, Ballabeni P, Niquille A. Effects of an interprofessional Quality Circle-Deprescribing Module (QC-DeMo) in Swiss nursing homes: a randomised controlled trial. BMC Geriatr. 2021 May 1;21(1):289. doi: 10.1186/s12877-021-02220-y. PMID 33933030
- [Derived] Cateau D, Ballabeni P, Mena S, Bugnon O, Niquille A. Deprescribing in nursing homes: Protocol for nested, randomised controlled hybrid trials of deprescribing interventions. Res Social Adm Pharm. 2021 Apr;17(4):786-794. doi: 10.1016/j.sapharm.2020.05.026. Epub 2020 May 27. PMID 32622774
- See also: Website of funding body — http://www.nfp74.ch/en/projects/in-patient-care/project-bugnon

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Nursing home
Period: Overall Study
Arm/Group | Intervention | Control
Started | NA; 27 Nursing home (No individual participants were recruited, only nursing homes.) | NA; 29 Nursing home (No individual participants were recruited, only nursing homes.)
Completed | NA; 27 Nursing home (No individual participants were recruited, only nursing homes.) | NA; 28 Nursing home (1 nursing home withdrew from the study. No individual participants were recruited, only nursing homes.)
Not Completed | NA; 0 Nursing home | NA; 1 Nursing home

BASELINE CHARACTERISTICS:
Population: The unit of analysis for the trial is the nursing home (NH); no individual NH residents were enroled. Therefore, no data on age and gender can be provided.
Units Other Than Participants: Nursing home
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | NA | NA | NA
Number analyzed (Nursing home) | 27 | 29 | 56
Age, Customized [Count of Units; unit: Nursing home]
  n/a | NA — No individual NH residents were enroled. Therefore, no data on age and gender can be provided. | NA — No individual NH residents were enroled. Therefore, no data on age and gender can be provided. | NA — Total not calculated because data are not available (NA) in one or more arms.
Sex/Gender, Customized [Count of Units; unit: Nursing home]
  n/a | NA — No individual NH residents were enroled. Therefore, no data on age and gender can be provided. | NA — No individual NH residents were enroled. Therefore, no data on age and gender can be provided. | NA — Total not calculated because data are not available (NA) in one or more arms.
Race/Ethnicity, Customized [Count of Units; unit: Nursing home]
  n/a | NA — No individual NH residents were enroled. Therefore, no data on ethnicity can be provided. | NA — No individual NH residents were enroled. Therefore, no data on ethnicity can be provided. | NA — Total not calculated because data are not available (NA) in one or more arms.
Region of Enrollment [Number; unit: participants]
  Switzerland | 27 | 29 | 56
NH mission [Count of Units; unit: Nursing home] — Psycho-geriatric mission include NHs with mixed mission (both geriatric and psycho-geriatric)
  Nursing home
    Geriatric | 16 | 20 | 36
    Psycho-geriatric | 11 | 9 | 20
Number of average residents [Median (Inter-Quartile Range); unit: Number of average residents] — Total number of days spent in the nursing home (NH) by all residents in a year, divided by 365. Roughly equivalent to the number of beds in the NH, but accounting for "empty beds".
  NOT equivalent to the average number of residents, as this measure would require the knowledge of individual residents, which was not collected for this study. Only data at the NH level (e.g. total number of days spent in the H) were collected.
  Number of average residents | 48 [33 to 81] | 35 [22 to 47] | 43 [23 to 62]
Percentage of potentially inappropriate galenic units [Median (Inter-Quartile Range); unit: percent] — Percentage of potentially inappropriate galenic units, relative to the total number of galenic units used in the nursing home in a year.
  percent | 26 [20 to 30] | 22 [6 to 45] | 24 [18 to 29]
Overall number of potentially inappropriate DDD [Median (Inter-Quartile Range); unit: DDD per average resident and per day] — Potentially inappropriate medications are classified as "to avoid" (indicating that inappropriate use is more likely) or "to reevaluate". The overall number is the sum of these two categories.
  DDD per average resident and per day | 2.4 [1.8 to 2.7] | 2.4 [1.9 to 2.7] | 2.4 [1.8 to 2.7]
Number of potentially inappropriate DDD to avoid [Median (Inter-Quartile Range); unit: DDD per average resident and per day] — Potentially inappropriate medications are classified as "to avoid" (indicating that inappropriate use is more likely) or "to reevaluate".
  DDD per average resident and per day | 0.3 [0.2 to 0.5] | 0.4 [0.2 to 0.5] | 0.4 [0.2 to 0.5]
Number of potentially inappropriate DDD to reevaluate [Median (Inter-Quartile Range); unit: DDD per average resident and per day] — Potentially inappropriate medications are classified as "to avoid" (indicating that inappropriate use is more likely) or "to reevaluate".
  DDD per average resident and per day | 1.9 [1.6 to 2.3] | 2.1 [1.6 to 2.3] | 2.0 [1.6 to 2.3]
Mortality rate [Median (Inter-Quartile Range); unit: percent] — Percentage of residents in the nursing home (NH) having died in the considered year, relative to the total number of residents having stayed at the NH during this year.
  percent | 32 [26 to 42] | 34 [26 to 48] | 34 [26 to 43]
Days in hospital [Median (Inter-Quartile Range); unit: Days] — Total number of days spent in the hospital by all nursing residents in the considered year, divided by the number of average residents.
  Days | 2.7 [1.5 to 3.4] | 2.5 [1.5 to 3.8] | 2.5 [1.5 to 3.4]
Number of falls [Median (Inter-Quartile Range); unit: Falls per avg. resident and per year] — Total number of falls that occured in the nursing home during the considered year, divided by the number of average residents.
  Falls per avg. resident and per year | 2.3 [1.7 to 3.3] | 2.3 [1.4 to 3.1] | 2.3 [1.5 to 3.2]
Rate of physical restraints use [Median (Inter-Quartile Range); unit: Percent] — Percentage of residents in the nursing home (NH) with at least one day with physical restraints during the considered year, relative to the total number of residents having stayed at the NH during this year.
  Percent | 23 [12 to 39] | 27 [12 to 45] | 24 [12 to 43]

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Potentially Inappropriate Galenic Units
Description: The primary outcome is the percentage, at follow-up, of potentially inappropriate galenic units at follow-up, relative to the total number of galenic units used in the nursing home.
Time Frame: 12 months
Population: The analysis level is the nursing home; no data on individual residents were collected
Measure: Mean (Standard Deviation); unit: percent
Units Other Than Participants: Nursing homes
Arm/Group | Intervention | Control
Number analyzed (Participants) | NA | NA
Number analyzed (Nursing homes) | 27 | 28
percent | 24 (7) | 23 (9)
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p < 0.05, Regression, Linear; Dependant variable = follow-up value; adjusted for baseline value, canton, avg number of residents, mission; Slope = -1.4, 95% CI 2-sided [-3.8 to 1.0]

2. Primary Outcome: Number of Potentially Inappropriate Defined Daily Doses (DDDs) Per Average Resident and Per Day
Description: Sum of Defined Daily Doses identified as potentially inappropriate (PIM, see protocol for assessement method), divided by the total number of days spent in the NH
Time Frame: 12 months
Population: The analysis level is the nursing home; no data on individual residents were collected
Measure: Mean (Standard Deviation); unit: PIM DDD per avg resident per day
Units Other Than Participants: Nursing homes
Arm/Group | Intervention | Control
Number analyzed (Participants) | NA | NA
Number analyzed (Nursing homes) | 27 | 28
PIM DDD per avg resident per day | 2.1 (0.5) | 2.3 (0.5)
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p < 0.05, Regression, Linear; Dependant variable = number of PIM DDD at follow-up, adjusted for baseline value, canton, avg number of residents, mission; Slope = -0.18, 95% CI 2-sided [-0.39 to 0.03]

3. Secondary Outcome: Number of Potentially Inappropriate DDD to Avoid
Description: Sum of Defined Daily Doses identified as "to avoid" (see protocol for assessement method), divided by the total number of days spent in the NH.
Time Frame: 12 months
Population: The analysis level is the nursing home; no data on individual residents were collected
Measure: Mean (Standard Deviation); unit: Number of PIM DDD per avg resident
Units Other Than Participants: Nursing homes
Arm/Group | Intervention | Control
Number analyzed (Participants) | NA | NA
Number analyzed (Nursing homes) | 27 | 28
Number of PIM DDD per avg resident | 0.3 (0.2) | 0.3 (0.2)
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p < 0.05, Regression, Linear; [statistical method as in outcome 2, analysis 1]; Slope = -0.035, 95% CI 2-sided [-0.095 to 0.025]

4. Secondary Outcome: Number of Potentially Inappropriate DDD to Reevaluate
Description: Sum of Defined Daily Doses identified as "to reevaluate" (see protocol for assessement method), divided by the total number of days spent in the NH.
Time Frame: 12 months
Population: The analysis level is the nursing home; no data on individual residents were collected
Measure: Mean (Standard Deviation); unit: Number of PIM DDD per avg resident
Units Other Than Participants: Nursing homes
Arm/Group | Intervention | Control
Number analyzed (Participants) | NA | NA
Number analyzed (Nursing homes) | 27 | 28
Number of PIM DDD per avg resident | 1.8 (0.5) | 2.0 (0.5)
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p < 0.05, Regression, Linear; [statistical method as in outcome 2, analysis 1]; Slope = -0.237, 95% CI 2-sided [-0.435 to -0.040]

5. Secondary Outcome: Number of Hospital Days
Description: The number of days spent in the hospital by average resident
Time Frame: 12 months
Population: The analysis level is the nursing home; no data on individual residents were collected
Measure: Mean (Standard Deviation); unit: Days per avg resident and per year
Units Other Than Participants: Nursing homes
Arm/Group | Intervention | Control
Number analyzed (Participants) | NA | NA
Number analyzed (Nursing homes) | 24 | 27
Days per avg resident and per year | 3.1 (1.5) | 2.5 (1.7)
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p < 0.05, Regression, Linear; Dependent variable = follow-up value, adjusted for baseline value, canton, avg number of residents, interaction between mission and group; Slope = 1.55, 95% CI 2-sided [0.164 to 2.938]

6. Secondary Outcome: Mortality Rate
Description: Number of residents of the nursing home having died during the considered year, divided by the total number of residents having stayed in the nursing home.
Time Frame: 12 months
Population: The analysis level is the nursing home; no data on individual residents were collected
Measure: Mean (Standard Deviation); unit: Percent of residents having died
Units Other Than Participants: Nursing homes
Arm/Group | Intervention | Control
Number analyzed (Participants) | NA | NA
Number analyzed (Nursing homes) | 25 | 26
Percent of residents having died | 31 (14) | 38 (8)
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p < 0.05, Regression, Linear; [statistical method as in outcome 5, analysis 1]; Slope = -12.7, 95% CI 2-sided [-21.5 to -4.0]

7. Secondary Outcome: Number of Falls Per Average Resident and Per Year
Description: Number of falls per average resident and per year
Time Frame: 12 months
Population: The analysis level is the nursing home; no data on individual residents were collected.
Measure: Mean (Standard Deviation); unit: Falls per avg resident and per year
Units Other Than Participants: Nursing homes
Arm/Group | Intervention | Control
Number analyzed (Participants) | NA | NA
Number analyzed (Nursing homes) | 25 | 27
Falls per avg resident and per year | 3.0 (1.9) | 2.6 (1.1)
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p < 0.05, Regression, Linear; Dependent variable = follow-up value, adjusted for baseline value, canton, avg number of residents; Slope = -0.165, 95% CI 2-sided [-0.754 to 0.424]

8. Secondary Outcome: Percentage of Residents With at Least One Day of Physical Restraints Use
Description: Number of residents of the nursing home with at least one day of physical restraints use during the considered year, divided by the total number of residents having stayed in the nursing home.
Time Frame: 12 months
Population: The analysis level is the nursing home; no data on individual residents were collected.
Measure: Mean (Standard Deviation); unit: Proportion of res with phys restraints
Units Other Than Participants: Nursing homes
Arm/Group | Intervention | Control
Number analyzed (Participants) | NA | NA
Number analyzed (Nursing homes) | 25 | 27
Proportion of res with phys restraints | 33 (27) | 37 (23)
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p < 0.05, Regression, Linear; Dependent variable = follow-up value, adjusted for baseline value, canton, avg number of residents; Slope = -4.2, 95% CI 2-sided [-16.0 to 7.6]

ADVERSE EVENTS:
Description: Individual adverse events were not collected for this study; safety outcomes are included in the Outcomes section
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 921/2899 | 717/2113
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2020-02-05): https://cdn.clinicaltrials.gov/large-docs/42/NCT03688542/Prot_001.pdf
  • Statistical Analysis Plan (2018-08-07): https://cdn.clinicaltrials.gov/large-docs/42/NCT03688542/SAP_002.pdf